CLINICAL TRIAL: NCT06971627
Title: The Effect of Telehealth Monitoring on Medication Compliance, Self-Efficacy and Quality of Life in Patients With İnflammatory Bowel Disease
Brief Title: Telehealth Monitoring in Inflammatory Bowel Disease: Effects on Medication Compliance, Self-Efficacy, and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Zeliha Tülek, RN, MSc, PhD, Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Inflammatory Bowel Disease
Record Dates: First submitted 2025-05-07; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Disease (IBD); Medication Compliance; Quality of Life; Telehealth Monitoring
Keywords: Inflammatory Bowel Disease; Medication Compliance; Self-Efficacy; Quality of Life; Telehealth Monitoring; Crohn's Disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Medication Adherence; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomized controlled trial with a pretest-posttest design, consisting of two groups: an intervention group and a control group.
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will be included in a structured telehealth monitoring program led by a nurse for 12 weeks.
  Interventions: Behavioral: Nurse-led Telehealth Monitoring Program
- Control group (Other): Participants in the control group will only receive standard care. No additional interventions will be implemented during the 12-week period.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Nurse-led Telehealth Monitoring Program — Participants in the intervention group will be included in a structured telehealth monitoring program led by a nurse for 12 weeks.
  Arms: Intervention Group
Other: No intervention — Participants in the control group will only receive standard care. No additional interventions will be implemented during the 12-week period.
  Arms: Control group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of nurse-led telehealth monitoring on medication adherence, self-efficacy, and quality of life in individuals with inflammatory bowel disease (IBD). The study will be conducted at the IBD Outpatient Clinic of Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty. Participants will be randomly assigned to either an intervention group receiving a 3-month structured telehealth program (including education, counseling, phone calls, and reminders) or a control group receiving only standard care and an educational booklet. Outcomes will be assessed at baseline and after 12 weeks.

DETAILED DESCRIPTION:
This randomized controlled trial aims to assess the impact of a nurse-led telehealth monitoring program on medication adherence, self-efficacy, and quality of life in patients with inflammatory bowel disease (IBD). The study will be conducted at the IBD Outpatient Clinic, Istanbul University-Cerrahpaşa, Cerrahpaşa Medical Faculty Hospital.

Participants will be randomly assigned to either an intervention or control group. The intervention group will receive a 12-week structured telehealth program including an educational booklet, video content, a Zoom-based group session, biweekly phone calls, and reminder messages. The control group will receive only standard care and the educational booklet, with no additional intervention.

Assessments will be conducted at baseline (Week 0) and at the end of the intervention (Week 12) using validated tools: Harvey-Bradshaw Index (HBI), Simple Clinical Colitis Activity Index (SCCAI), Medication Adherence Report Scale (MARS), MedTake Test, IBD Self-Efficacy Scale, IBD Quality of Life Questionnaire, and IBD Distress Scale.

The effectiveness of the intervention will be determined by comparing pre- and post-intervention outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* Individuals aged 18 years or older
* Able to read and write in Turkish
* Diagnosed with inflammatory bowel disease (IBD) for at least 6 months
* In clinical remission (Harvey-Bradshaw Index score < 5 or Simple Clinical Colitis Activity Index score < 3)
* Able to use a smartphone
* Have access to an online messaging application (e.g., WhatsApp) and a valid e-mail address
* Capable of downloading and using a mobile or computer-based video conferencing application (e.g., Zoom)
* Willing to participate in the study voluntarily

Exclusion Criteria:

* Diagnosed with any psychiatric or cognitive disorder
* Having any condition that impairs communication
* Pregnant women
* Patients receiving infusion-based treatment
* Having an advanced chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Medication Adherence Report Scale (MARS) scores | Baseline (Week 0) and 12 weeks (3 months) following telehealth monitoring.
  This scale assesses self-reported medication adherence behavior. The outcome will evaluate the change in MARS scores from baseline to week 12 to determine the impact of the telehealth intervention on adherence.

SECONDARY OUTCOMES:
Change in MedTake Test scores | Baseline (Week 0) and 12 weeks (3 months) following telehealth monitoring.
  The MedTake test evaluates patients' ability to understand and manage their oral medication regimen. This outcome will examine improvements in medication-taking skills from baseline to the end of the 12-week intervention.
Change in Harvey-Bradshaw Index scores (for Crohn's Disease) and Change in Simple Clinical Colitis Activity Index scores (for Ulcerative Colitis) | Baseline (Week 0) and 12 weeks (3 months) following telehealth monitoring
  These indices measure disease activity in Crohn's Disease and Ulcerative Colitis, respectively. The outcome will track changes in disease activity from baseline to week 12 following the telehealth monitoring.
Change in Inflammatory Bowel Disease (IBD) Self-Efficacy Scale scores | Baseline (Week 0) and 12 weeks (3 months) following telehealth monitoring.
  This scale measures a patient's confidence in managing their IBD-related health challenges. The outcome will assess changes in self-efficacy levels between baseline and week 12.
Change in Inflammatory Bowel Disease Questionnaire scores | Baseline (Week 0) and 12 weeks (3 months) following telehealth monitoring.
  This questionnaire evaluates the quality of life in patients with IBD. The outcome will assess the effect of the intervention on quality of life by comparing scores at baseline and after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kimya Kılıçaslan, PhD Candidate, Principal Investigator — Istanbul University - Cerrahpasa Institute of Graudate Studies; Zeliha Tulek, PhD, Prof., Study Director — Istanbul University - Cerrahpasa, Florence Nightingale Faculty of Nursing; Aykut Ferhat Çelik, MD, Prof., Study Chair — Istanbul University - Cerrahpasa Cerrahpaşa Faculty of Medicine Department of Gastroenterology
Locations (1):
- Istanbul University - Cerrahpasa Cerrahpaşa Faculty of Medicine Department of Gastroenterology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon M, Sinopoulou V, Lakunina S, Gjuladin-Hellon T, Bracewell K, Akobeng AK. Remote care through telehealth for people with inflammatory bowel disease. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014821. doi: 10.1002/14651858.CD014821.pub2. PMID 37140025
- [Background] Pang L, Liu H, Liu Z, Tan J, Zhou LY, Qiu Y, Lin X, He J, Li X, Lin S, Ghosh S, Mao R, Chen M. Role of Telemedicine in Inflammatory Bowel Disease: Systematic Review and Meta-analysis of Randomized Controlled Trials. J Med Internet Res. 2022 Mar 24;24(3):e28978. doi: 10.2196/28978. PMID 35323120